CLINICAL TRIAL: NCT01824771
Title: Effects of Continuous Veno-venous Haemofiltration on Plasma Lactate in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liu Yong-Jun, Doctor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 2013232
Record Dates: First submitted 2013-03-28; First posted 2013-04-05 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Kidney Injury, Acute
Keywords: Continuous veno-venoous haemofiltration; Plasma lactate; Critical illness; Acute kidney injurytissue perfusion; Multiple organ dysfunction syndrome
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Plasma lactate were measured — Three different doses (20 ml/kg/h, 35 ml/kg/h and 45 ml/kg/h) of CVVH were applied to critically ill patients who experiencing CVVH. Each dose of CVVH was sequentially gave to each patient and lasted for 30 minutes separately

SUMMARY:
Continuous Veno-Venous Hemofiltration (CVVH) can eliminate metabolic products effectively and replace renal function partly. It is widely used in intensive care units (ICUs), especially for patients with acute kidney injury/failure in an unstable hemodynamic status. Lactate is a molecule smaller than glucose, which can pass through filtration membrane freely in CVVH. Therefore, the blood lactate concentrations would no longer reflect tissue oxygenation status in patients with unstable hemodynamic status. However, there is no prospective study evaluated the effect of CVVH on lactate removal in critically ill patients. The influence of different dose of CVVH on lactate elimination is not clear in patients with different level of serum lactate. Our study aimed to find out how the dose of CVVH effects on lactate clearance, and then re-estimate the prognostic value of lactate in critically ill patients with CVVH.

ELIGIBILITY:
Inclusion Criteria:

1. The critical ill patients with acute kidney injury
2. Patients requiring continuous veno-venous hemofiltration
3. APACHE II scores more than 12
4. Arterial lactate is higher than 0.5mmol/L but lower than 15mmol/L (due to the sensitivity and optimal measuring range of the equipment)
5. Continuous veno-venous hemofiltration for at least 12 hrs
6. Hemo-filter age of <24 hrs

Exclusion Criteria:

1. APACHE II scores lower than 12
2. patients' age are more than 75Y or lower than 18Y

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was carried out in Surgical Intensive Care Unit (SICU) of the first affiliated hospital, Sun Yat-sen University.The project has been approved by Ethics Committee of Sun Yat-sen University. All the subjects have signed written informed consent.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-03-03 (Actual); Primary Completion 2015-03-03 (Actual); Study Completion 2015-03-20 (Actual)

PRIMARY OUTCOMES:
plasma lactate | 30 minutes
  Each dose of CVVH was lasted for 30 minutes separately. Blood samples were draw pre-(A) and post-dialyzer (V) site after each dosage of CVVH was carried out for 30 minutes and then plasma lactates were measured immediately

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Levraut J, Ciebiera JP, Jambou P, Ichai C, Labib Y, Grimaud D. Effect of continuous venovenous hemofiltration with dialysis on lactate clearance in critically ill patients. Crit Care Med. 1997 Jan;25(1):58-62. doi: 10.1097/00003246-199701000-00013. PMID 8989177